CLINICAL TRIAL: NCT01997892
Title: TRANSFORM - Observational Cohort Study of Aranesp Use in EU Haemodialysis Patients Switched From Mircera
Brief Title: TRANSFORM - Observational Cohort Study of Darbepoetin Alfa Use in European Union (EU) Hemodialysis Patients Switched From PEG Epoetin Beta
Acronym: TRANSFORM
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120126
Record Dates: First submitted 2012-12-18; First posted 2013-11-28 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Anemia
Keywords: CKD; Darbepoetin Alfa; Dialysis; Hemodialysis; Anemia; Peg epoetin beta
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease (CKD): Participants with CKD on dialysis and treated with PEG epoetin beta for a minimum of 14 weeks immediately prior to being switched to darbepoetin alfa.

SUMMARY:
To describe the time course of hemoglobin concentration in EU hemodialysis patients switched from methoxy polyethylene glycol-epoetin beta (PEG epoetin beta; Mircera) to darbepoetin alfa (Aranesp).

DETAILED DESCRIPTION:
This is a multi-centre, observational cohort study of EU hemodialysis patients whose erythropoiesis stimulating agent (ESA) therapy has been switched from PEG epoetin beta to darbepoetin alfa. Data will be collected for the period spanning 14 weeks prior to switch through to 26 weeks post-switch.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age. CKD diagnosis, receiving hemodialysis
* Received PEG epoetin beta for 14weeks prior to switching to darbepoetin alfa and received at least one dose of darbepoetin alfa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD dialysed patients from EU centers treated with PEG epoetin beta for a minimum of 14weeks prior to switching to darbepoetin alfa.
Sampling Method: Non-Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (29):
- Research Site, Edegem, Belgium
- France (21):
  - Research Site, Antony
  - Research Site, Aurillac
  - Research Site, Béziers
  - Research Site, Blois
  - Research Site, Boulogne-sur-Mer
  - Research Site, Cahors
  - Research Site, Essey-lès-Nancy
  - Research Site, Grabels
  - Research Site, La Réunion
  - Research Site, La Roche-sur-Yon
  - Research Site, Libourne
  - Research Site, Lille
  - Research Site, Metz
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Saint-Denis de La Réunion
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Pierre
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Vandœuvre-lès-Nancy
- Germany (2):
  - Research Site, Kiel
  - Research Site, Nordhorn
- Research Site, Athens, Greece
- Research Site, Arnhem, Netherlands
- Spain (2):
  - Research Site, Ribeira, Galicia
  - Research Site, Santiago de Compostela, Galicia
- Research Site, Sion, Switzerland

REFERENCES:
- [Derived] Donck J, Gonzalez-Tabares L, Chanliau J, Martin H, Stamatelou K, Manamley N, Farouk M, Addison J. Preservation of anemia control and weekly ESA dosage after conversion from PEG-Epoetin beta to darbepoetin alfa in adult hemodialysis patients: the TRANSFORM study. Adv Ther. 2014 Nov;31(11):1155-68. doi: 10.1007/s12325-014-0161-5. Epub 2014 Nov 1. PMID 25367412
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 28 August 2012; Last patient enrolled 3 July 2013.
Groups:
- Chronic Kidney Disease (CKD): Participants with CKD on dialysis and treated with PEGylated (PEG) epoetin beta immediately prior to being switched to darbepoetin alfa.
Period: Overall Study
Arm/Group | Chronic Kidney Disease (CKD)
Started | 1027
Received Darbepoetin Alfa | 987
Completed | 959
Not Completed | 68
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 6
Not completed — Death | 14
Not completed — Renal transplant | 8
Not completed — Other | 3
Not completed — Study completion data not recorded | 35

BASELINE CHARACTERISTICS:
Population: The Primary Analysis Set included all participants who received at least one dose of darbepoetin alfa who completed 26 weeks post-switch on darbepoetin alfa, did not receive another erythropoiesis stimulating agent during this period and had at least one hemoglobin value per month recorded for a minimum of any 4 months post-switch.
Groups:
- Chronic Kidney Disease (CKD): Participants with CKD on dialysis and treated with PEG epoetin beta immediately prior to being switched to darbepoetin alfa.
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 785
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 344
  Male | 441

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentration at Monthly Intervals
Description: Hemoglobin concentration from 3 months prior to switch to darbepoetin alfa until the end of the observation period.
Time Frame: Month -3, -2, -1 (pre-switch), and Month 1, 2, 3, 4, 5 and 6 (post-switch)
Population: Primary analysis set; participants with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 785
g/dL
  Month -3 (n=725) | 11.27 (1.09)
  Month -2 (n=766) | 11.26 (1.08)
  Month -1 (n=769) | 11.19 (1.06)
  Month 1 (n=763) | 11.14 (1.09)
  Month 2 (n=755) | 11.36 (1.13)
  Month 3 (n=749) | 11.48 (1.14)
  Month 4 (n=754) | 11.38 (1.15)
  Month 5 (n=739) | 11.33 (1.15)
  Month 6 (n=742) | 11.29 (1.14)

2. Secondary Outcome: PEG Epoetin Beta Dose From the Start of the Observation Period Until the Switch
Description: Mean weekly doses were calculated per participant by first calculating a mean daily dose for the interval (by dividing each dose evenly between the days bounded by its date of administration and the day before the next dose, then taking a mean of these partial doses for the days in the interval) and multiplying by 7 to convert to a weekly dose. Weekly doses >150 μg have been excluded as they were deemed infeasible values derived by the algorithm.
Time Frame: Month -3, Month -2, Month -1
Population: Primary analysis set; participants with available data at each time point (indicated by "n").
Measure: Geometric Mean (95% Confidence Interval); unit: μg/week
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 785
μg/week
  Month -3 (n=740) | 27.7 (23.7) [26.3 to 29.2]
  Month -2 (n=779) | 26.5 (22.1) [25.2 to 27.9]
  Month -1 (n=783) | 27.4 (24.2) [26.0 to 28.8]

3. Secondary Outcome: Darbepoetin Alfa Dose From the Switch Date Until the End of the Observation Period
Description: as for outcome 2
Time Frame: Month 1, 2, 3, 4, 5 and 6
Population: Primary analysis set; participants with available data at each time point (as indicated by "n").
Measure: Geometric Mean (95% Confidence Interval); unit: μg/week
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 785
μg/week
  Month 1 (n=782) | 29.4 (26.1) [27.9 to 30.9]
  Month 2 (n=778) | 27.8 (26.0) [26.3 to 29.3]
  Month 3 (n=780) | 25.4 (26.8) [23.9 to 27.0]
  Month 4 (n=779) | 23.3 (27.6) [21.9 to 24.9]
  Month 5 (n=777) | 23.8 (26.5) [22.3 to 25.3]
  Month 6 (n=769) | 25.6 (25.5) [24.1 to 27.1]

4. Secondary Outcome: Dose Ratio Measured at the Time of Switch From PEG Epoetin Beta to Darbepoetin Alfa
Description: Dose ratio is the average weekly dose of the first darbepoetin alfa dose divided by the average weekly dose of peg-epoetin beta at switch (μg darbepoetin alfa per 1 μg pegylated-epoetin beta).
Time Frame: Week -1 and Week 1
Population: Primary analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Chronic Kidney Disease (CKD)
Number analyzed (Participants) | 785
ratio | 1.06 [1.01 to 1.11]

5. Secondary Outcome: Hemoglobin Concentration Rate of Change by Period
Description: The hemoglobin rate of change is the maximum monthly increase and maximum monthly decrease for the pre- and post-switch periods. Within each period, the difference was calculated between each hemoglobin value and the most recent hemoglobin value taken at least 28 days previously. The rate of change was calculated by dividing this difference by the number of days in the interval and multiplying by 28. The maximum and minimum rate of change was then determined per participant.
Time Frame: Thre months prior to switch and 6 months after the switch
Population: Primary Analysis Set with available data
Measure: Mean (Standard Deviation); unit: g/dL/4 week
Groups:
- Pre-switch Period: From 3 months prior to the switch until the date of the switch to darbepoetin alfa.
- Post-switch Period: From the date of the switch to darbepoetin alfa, until up to 6 months.
Arm/Group | Pre-switch Period | Post-switch Period
Number analyzed (Participants) | 774 | 785
g/dL/4 week
  Highest change during period | 0.64 (0.71) | 1.17 (0.74)
  Lowest change during period | -0.73 (0.86) | -1.21 (0.88)

6. Secondary Outcome: Percentage of Participants With Hemoglobin Excursions
Description: The percentage of participants with at least one hemoglobin excursion, defined as hemoglobin concentrations below 10.0 g/dL and above 12.0 g/dL during the pre- and post-switch periods.
Time Frame: Month -3, -2, -1, 1, 2, 3, 4, 5 and 6
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Excursions <10.0 g/dL: Hemoglobin excursions below 10.0 g/dL
- Excursions > 12.0 g/dL: Hemoglobin excursions above 12.0 g/dL
Arm/Group | Excursions <10.0 g/dL | Excursions > 12.0 g/dL
Number analyzed (Participants) | 785 | 785
percentage of participants
  Month -3 | 16.8 [14.3 to 19.6] | 29.0 [25.9 to 32.4]
  Month -2 | 17.7 [15.1 to 20.6] | 29.0 [25.9 to 32.4]
  Month -1 | 15.7 [13.2 to 18.4] | 24.8 [21.9 to 28.0]
  Month 1 | 17.8 [15.2 to 20.7] | 23.1 [20.2 to 26.2]
  Month 2 | 13.6 [11.3 to 16.2] | 29.3 [26.1 to 32.6]
  Month 3 | 11.7 [9.6 to 14.2] | 33.1 [29.8 to 36.5]
  Month 4 | 13.8 [11.4 to 16.4] | 32.6 [29.3 to 36.0]
  Month 5 | 12.2 [10.0 to 14.7] | 27.8 [24.7 to 31.0]
  Month 6 | 14.6 [12.2 to 17.3] | 26.5 [23.4 to 29.7]

ADVERSE EVENTS:
Time Frame: The observation period for individual participants spanned 14 weeks prior to switching from PEG epoetin beta to darbepoetin alfa to a maximum of 26 weeks post-switch.
Description: Adverse drug reactions in the Full Analysis Set (all eligible enrolled participants who received at least one dose of darbepoetin alfa) are reported.
Arm/Group | Pre-switch Period | Post-switch Period
Serious Adverse Events (participants affected / at risk) | 0/987 | 0/987
Other Adverse Events (participants affected / at risk) | 0/987 | 1/987
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-switch Period (N=987) | Post-switch Period (N=987)
Hot flush (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.